CLINICAL TRIAL: NCT03937284
Title: Lipoprotein Lipidic Composition, Lipopolysaccharide Binding Protein, and Bacterial Endotoxin Exposure in Parkinson's Disease: A Pilot Study
Brief Title: Lipoprotein Metabolism and Bacterial Lipopolysaccharide in Parkinson's Disease
Acronym: LiMBaLiP
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Collaborators: Istituti Clinici di Perfezionamento di Milano (Other)
Responsible Party: Principal Investigator, roberta cazzola, Principal Investigator, University of Milan
Other Study IDs: Unimi
Record Dates: First submitted 2019-04-16; First posted 2019-05-03 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Parkinson Disease
Keywords: Lipoproteins; Lipopolysaccharide; Lipopolysaccharide binding protein; Inflammation
MeSH Terms: conditions — Parkinson Disease; Inflammation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma and erythrocytes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parkinson's patients: Patients with Parkinson disease evaluated in agreement with UK Brain Bank criteria
  Interventions: Other: Patients not treated
- Control group: Subject matched for sex, age and BMI
  Interventions: Other: Patients not treated

INTERVENTIONS:
Other: Patients not treated

SUMMARY:
Patients with Parkinson's disease (PD) present an impaired intestinal permeability with consequent lipopolysaccharide (LPS) translocation in the systemic circulation. Plasmatic lipoproteins play a key role in the detoxification of LPS.

The investigators aim to study the relationships between lipoprotein chemical composition and plasma LPS circulation in PD.

DETAILED DESCRIPTION:
Bacterial lipopolysaccharides are able to produce neuroinflammation and dopaminergic receptors degeneration. In addition, they may produce an accumulation of α-synuclein in the area of the substantia Nigra. Recent studies have shown that α-synuclein aggregates may be present also in gastrointestinal neurons of patients with PD. This last finding led to the hypothesis that the intestine might be an early site of PD disease in response to an environmental toxin or pathogen. Forsyth et al. have discovered an impaired intestinal permeability in subjects with recently diagnosed PD, and they found positive correlations between this factor, exposure to LPS and alpha-synuclein accumulation in gastrointestinal neurons. Plasma lipoproteins play a key role in the detoxification of bacterial endotoxins. Lipoprotein chemical composition is related to their detoxing properties. To the best of investigator knowledge, the relationships between lipoprotein chemical composition and LPS in PD have not yet been investigated. Therefore, the aims of this study are: I) to evaluate the chemical composition of VLDL, LDL and HDL in subjects with PD compared to a control group; 2) to analyze the activity of plasma lipid transfer proteins and LPS plasma levels in the same groups of subjects; III) finally, to investigate the correlations between the analyzed parameters.

Subjects and method Twenty patients with PD and twenty healthy controls were recruited for the study. Fasting blood samples were taken for routine laboratory analysis and for the separation of EDTA plasma. Plasma samples stored at -80°C until were used for lipoprotein isolation and analysis and for the measurement of lipid transfer protein and LPS levels.

ELIGIBILITY:
Parkinson's patients

Inclusion Criteria:

* Diagnosis of Parkinson disease in agreement with UK Brain Bank
* Farmacological treatment with L-Dopa and/or dopaminergic agonist or diagnosis de novo
* BMI 18.5 - 29.9 kg/m^2
* Informed consent signature

Exclusion criteria:

* Presence of type 1 and type 2 diabetes mellitus
* Presence of major chronic diseases of the digestive tract.
* Pregnancy in progress
* Subjects subjected to antihypertensive therapies or statins or with drugs that can change metabolic status and insulin sensitivity (e.g. chronic oral steroid therapy)
* Subjects affected by endocrine pathologies (e.g. Cushing disease, uncontrolled thyroid disease)
* Presence of known renal insufficiency or creatinine levels greater than 1.8 mg/dl
* Presence of chronic liver disease or ALT and AST levels exceeding two standard deviations from normal levels
* Presence of malignant disease
* Alcohol or drug abuse
* Major psychiatric disorders
* Subjects dedicated to intense and agonistic physical activity.

Control group

Inclusion criteria

* Absence of major disease
* BMI 18.5 - 29.9 kg/m^2
* Informed consent signature

Exclusion Criteria:

* Presence of type 1 and type 2 diabetes mellitus
* Presence of major chronic diseases of the digestive tract.
* Pregnancy in progress
* Subjects subjected to antihypertensive therapies or statins or with drugs that can change metabolic status and insulin sensitivity (e.g. chronic oral steroid therapy)
* Subjects affected by endocrine pathologies (e.g. Cushing disease, uncontrolled thyroid disease)
* Presence of known renal insufficiency or creatinine levels greater than 1.8 mg/dl
* Presence of chronic liver disease or ALT and AST levels exceeding two standard deviations from normal levels
* Presence of malignant disease
* Alcohol or drug abuse
* Major psychiatric disorders
* Subjects dedicated to intense and agonistic physical activity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parkinson affected patients and healthy controls matched for sex, age and BMI in agreement with inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2016-05-03 (Actual); Primary Completion 2017-10-20 (Actual); Study Completion 2017-10-20 (Actual)

PRIMARY OUTCOMES:
LPS | through study completion an average of 1 year
  LPS plasma levels (EU/L)
Lipoprotein chemical composition | through study completion an average of 1 year
  Cholesterol (mg/dL); HDL-cholesterol (mg/dL); triglycerides (mg/dL); phospholipids (mg/dL), apoproteins (mg/dL) of VLDL, LDL and HDL

SECONDARY OUTCOMES:
Plasma lipid transfer proteins | through study completion an average of 1 year
  Lipopolysaccharide binding protein (ng/mL), cholesterol ester transfer protein (ng/mL), phospholipid transfer protein (ng/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Cazzola, PhD, Principal Investigator — University of Milan
Locations (1):
- ASST Centro Specialistico Ortopedico Traumatologico Gaetano Pini-CTO, Milan, Italy

REFERENCES:
- [Background] Forsyth CB, Shannon KM, Kordower JH, Voigt RM, Shaikh M, Jaglin JA, Estes JD, Dodiya HB, Keshavarzian A. Increased intestinal permeability correlates with sigmoid mucosa alpha-synuclein staining and endotoxin exposure markers in early Parkinson's disease. PLoS One. 2011;6(12):e28032. doi: 10.1371/journal.pone.0028032. Epub 2011 Dec 1. PMID 22145021
- [Background] Lebouvier T, Chaumette T, Paillusson S, Duyckaerts C, Bruley des Varannes S, Neunlist M, Derkinderen P. The second brain and Parkinson's disease. Eur J Neurosci. 2009 Sep;30(5):735-41. doi: 10.1111/j.1460-9568.2009.06873.x. Epub 2009 Aug 27. PMID 19712093
- [Background] Han R. Plasma lipoproteins are important components of the immune system. Microbiol Immunol. 2010 Apr;54(4):246-53. doi: 10.1111/j.1348-0421.2010.00203.x. PMID 20377753
- [Background] Levels JH, Marquart JA, Abraham PR, van den Ende AE, Molhuizen HO, van Deventer SJ, Meijers JC. Lipopolysaccharide is transferred from high-density to low-density lipoproteins by lipopolysaccharide-binding protein and phospholipid transfer protein. Infect Immun. 2005 Apr;73(4):2321-6. doi: 10.1128/IAI.73.4.2321-2326.2005. PMID 15784577
- [Background] Hughes AJ, Ben-Shlomo Y, Daniel SE, Lees AJ. What features improve the accuracy of clinical diagnosis in Parkinson's disease: a clinicopathologic study. 1992. Neurology. 2001 Nov;57(10 Suppl 3):S34-8. No abstract available. PMID 11775598